CLINICAL TRIAL: NCT02325947
Title: A Multicentre Randomized Single Blind Placebo Controlled Study to Assess Efficacy of Hand Exoskeleton Controlled by Motor Imagery Based BCI for Post Stroke Patients Movement Rehabilitation
Brief Title: Efficacy of Hand Exoskeleton Controlled by BCI in Post Stroke Patients
Acronym: iMove
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Russian Academy of Medical Sciences (Other)
Collaborators: Pirogov Russian National Research Medical University (Other)
Responsible Party: Principal Investigator, Roman Lyukmanov, Research scientist, Russian Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: iMove
Record Dates: First submitted 2014-12-08; First posted 2014-12-25 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Poststroke/CVA Paresis
Keywords: Post stroke hand paresis brain injury
MeSH Terms: interventions — Brain-Computer Interfaces

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group (Experimental): Hand exoskeleton, brain-computer interface (BCI) 10 sessions of 45-minutes
  Interventions: Device: hand exoskeleton, brain-computer interface (BCI),
- Placebo group (Sham Comparator): Hand exoskeleton, sham BCI 10 sessions of 45-minutes (BCI imitation)
  Interventions: Device: hand exoskeleton, sham BCI

INTERVENTIONS:
Device: hand exoskeleton, brain-computer interface (BCI), — Hand exoskeleton, brain-computer interface (BCI) 10 sessions of 45-minutes
  Other Names: mind-machine interface
  Arms: Study group
Device: hand exoskeleton, sham BCI — Hand exoskeleton, sham BCI 10 sessions of 45-minutes (BCI imitation)
  Arms: Placebo group

SUMMARY:
The purpose of this study is to assess the efficacy of non-invasive BCI-exoskeleton technology based on EEG patterns recognition matching to motor imagery in post-stroke patients with hand paresis.

DETAILED DESCRIPTION:
The BCI training is based on EEG activity patterns recording during hand motor imagery. A subject sit comfortably 1m from a computer screen which presents visual instructions during the session. The robotic exoskeleton is fixed to the paretic hand. Subject visually fixate on a circle presented in the center of the screen and receive instructions from three surrounding rhomboidal arrows. Subject is given three commands instructing them to relax or imagine slow hand opening movement with the right or left hand. The "Relax" command means that the subject have to sit still and look at the center of the screen. Commands are presented randomly, each of 10 sec duration.

A visual cue provides the subject with feedback regarding the mental task recognition: the central circle turned green if the classifier recognizes the task in agreement with the given command, or remains white if the signal is not recognized. In addition to visual feedback the subject is provided with kinesthetic feedback: the exoskeleton is opening the hand when the classifier recognizes the imagery of paretic hand movement.

The EEG is registered with 30 electrodes distributed over the head in accordance with the standard international 10-20 system. EEG signals are filtered from 5-30Hz. A Bayesian approach for EEG pattern classifying is used in the system. The activity sources most relevant for BCI functioning will be identified using an independent component analysis (ICA). Classification accuracy will by measured with Cohen's kappa (Kohavi and Provost, 1998). The procedure may consist from up to three sessions, the duration of 1 session is 10 min, there are 5 min time brake between session and total duration of procedure is up to 45 min. The number of procedures - at least 10. The maximal interval between procedures is 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Medical history of primary acute cerebrovascular event (ischemic or hemorrhagic stroke) at least 4 weeks before screening
* focal stroke located in a hemisphere
* post stroke hand paresis (mild to plegia according to Medical Research Council (MRC) Scale for Muscle Strength)

Exclusion Criteria:

* Montreal Cognitive Assessment (MoCA) scale < 22
* Left handedness
* Sensory aphasia
* Severe impairment of vision
* Modified Ashworth Scale (MAS) ≥ 4

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-01; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in hand paresis level and hand muscle spasticity | Week 2
  ARAT; Fugl-Meyer, Modified Ashworth scale

SECONDARY OUTCOMES:
Long-term changes from Baseline in hand paresis level and hand muscle spasticity | week 4, week 12, week 24
  ARAT; Fugl-Meyer, Modified Ashworth scale

CONTACTS AND LOCATIONS:
Overall Officials: Roman Lyukmanov, MD, Principal Investigator — Russian Academy of Medical Sciences
Locations (1):
- Research Center of Neurology of RAMS, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Post-stroke Rehabilitation Training with a Motor-Imagery-Based Brain-Computer Interface (BCI)-Controlled Hand Exoskeleton: A Randomized Controlled Multicenter Trial — https://www.frontiersin.org/articles/10.3389/fnins.2017.00400/full